CLINICAL TRIAL: NCT03480035
Title: Ideal Point of Transluminal Light in Tracheal Intubation With a Light Wand
Status: Completed | Type: Observational
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Jiwon Lee, assistant professor, Keimyung University Dongsan Medical Center
Other Study IDs: lightwand intubation
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Neck Disease; Trismus; Tooth Abnormalities
MeSH Terms: conditions — Trismus; Tooth Abnormalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: lightwand intubation — intubation using lightwand

SUMMARY:
If the patients's teeth are weak or the mouth dose not open well, the lightwand is a useful device when endotracheal intubation is necessary.

Therefore, if the appropriate position of the light beam is determined and the distance of the light source suitable for intubation using the lightwand is obtained from anatomical structures such as thyroid cartilage and cricoid cartilage, it is clinically useful. Because it can prevent unnecessary deep insertion or shallow insertion that can cause damage to anatomical structures during intubation.

DETAILED DESCRIPTION:
Studies have been reported on the proper position to bend the lightwand and the appropriate angle to bend when performing endotracheal intubation with lightwand. For ease of procedure, the assistant has to lift the patient's lower jaw or perform a neck extension.

However, there is no report on the position of the lightbulb when the light passes through the front of the airway and neck and appears bright in the midpoint.

The prodcedure is as follows.

1. FOB examination and check position of light below 1cm from vocal cord
2. lightwand intubation aimed at checkpoint
3. measurement of distance from thyroid cartilage/cricoid cartilage to light point

ELIGIBILITY:
Inclusion Criteria:

* impossibility of neck extension
* trismus
* weak teeth

Exclusion Criteria:

* previous history of larynx or neck surgery
* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an adult patient who is 18 years of age or older who undergoes general anesthesia requiring intubation.
  Among them, patients who are unable to extend their necks, have trismus or have weak teeth are selected.
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
distance from lightbeam of the FOB to thyroid cartilage | before intubation
  we will measure straight distance from lightbeam of the FOB to thyroid cartilage on the surface of patient's neck
distance from lightbeam of the FOB to cricoid cartilage | before intubation
  we will measure straight distance from lightbeam of the FOB to cricoid cartilage on the surface of patient's neck

SECONDARY OUTCOMES:
distance from lightbeam of the FOB to sternal notch | before intubation
  we will measure straight distance from lightbeam of the FOB to sternal notch on the surface of patient's neck

CONTACTS AND LOCATIONS:
Overall Officials: Jiwon Lee, Dr., Principal Investigator — Dongsan Medical Center
Locations (1):
- Dongsan medical center, Daegu, South Korea

REFERENCES:
- [Derived] Cho E, Kim HC, Lee JM, Park JH, Ha N, Hong JH, Lee J. Evaluation of transmitted glow point at a priori chosen depth (1 cm below vocal cords) for lightwand intubation: a prospective observational study. J Int Med Res. 2020 Dec;48(12):300060520974249. doi: 10.1177/0300060520974249. PMID 33284717